CLINICAL TRIAL: NCT01675687
Title: Effects on Self-efficacy, Sustainability and Drop Out Rate Using Web Based Follow up Intervention in Obesity Treatment for Women
Brief Title: Web Based Follow up Intervention in Obesity Treatment for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FEM Süd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-12-098-VK ID by EC Vienna
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: dietary habits and obesity; exercise habits and obesity; cognition and obesity
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet (Experimental): Participants of this intervention group get follow up support via Internet.
  They have access to new inputs biweekly consisting of
  * Thematic inputs and instructions (e.g. advice on shopping, cooking, regular exercise on daily routine, motivation and more)
  * assignments promoting self-awareness and introspection
  * spreadsheets promoting self-monitoring
  News and updates (e.g. recipes, gymnastic classes, meetings of self support groups and more) will be available each month.
  Tailored feedback of their behaviour will be given by documentation on spreadsheets.
  Interventions: Behavioral: Follow Up Support
- Printed Manual (Experimental): Participants of this intervention group get follow up support via a printed manual.
  The manual consist of all the same inputs as are available to the Internet follow up group.
  * Thematic inputs and instructions (e.g. advice on shopping, cooking, regular exercise on daily routine, motivation and more)
  * assignments promoting self-awareness and introspection
  * spreadsheets promoting self-monitoring
  All inputs will be given at once at the beginning of the follow up intervention, only news and updates (e.g. recipes, gymnastic classes, meetings of self support groups and more) will be sent per mail each month.
  There is no tailored feedback of their behaviour as the paper-pencil documentation on spreadsheets can't be monitored by the psychologists.
  Interventions: Behavioral: Follow Up Support

INTERVENTIONS:
Behavioral: Follow Up Support — inputs will be based on elements derived from cognitive behavioural therapy, acceptance and commitment therapy, mindfulness and awareness training

SUMMARY:
This study is designed to verify that web based follow up intervention after a classic multidisciplinary face-to-face obesity treatment will reinforced nutrition and exercise self-efficacy, improve drop out rate and advance sustainability after weight loss of obese women.

Research Questions and Hypotheses

* How does a web based follow up intervention change self-efficacy of women participating in an obesity intervention?
* How does a web based follow up intervention affect the drop out rate of women participating in an obesity intervention?
* How does a web based follow up intervention influence sustainability of women participating in an obesity intervention?

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-80
* BMI 30-40
* Internet access
* Motivation and psychological stability to stay in a long term obesity intervention
* No medical conditions prohibiting moderate physical exercise

Exclusion Criteria:

* Men
* Age under 18 years
* BMI under 30 and above 40
* No Internet access
* No motivation and psychological stability to stay in a long term obesity intervention
* Medical conditions prohibiting moderate physical exercise

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in nutrition- and exercise self-efficacy | Primary outcome measure is assessed at the beginning of the follow up support (baseline) and after 6 months (at completion of the follow up intervention by Internet or printed manual)
  Changes in nutrition- and exercise self-efficacy will be measured by scores in questionnaires for nutrition- and exercise self-efficacy (Sportbezogene Selbstwirksamkeitserwartung - Fuchs & Schwarzer, 1994 and Weight Efficacy Life-Style Questionnaire - Clark et al. 1991). A change of more than one standard deviation will be considered significant.

SECONDARY OUTCOMES:
Dropout rate | Secondary outcome measure is assessed at the beginning of the follow up support (baseline) and after 6 months (at completion of the follow up intervention by Internet or printed manual)
  The Dropout rate will be compared by the number of women available for the last meeting at the end of the follw up intervention.

OTHER OUTCOMES:
Sustainability of weight loss | Further outcome measure is assessed at the beginning of the follow up support (baseline) and after 6 months (at completion of the follow up intervention by Internet or printed manual)
  Sustainability will be measured in
  * percentage of women successfully stabilized weight (range of ± 2 kg based on Cooper et al. (2008)
  * percentage of women keeping the scores or impair no more than 1 standard deviation in their test results ("Ad Eva Testsystem zur Diagnostik und Evaluation bei Adipositas" - Ardelt-Gattinger und Meindl, 2009; "Sportbezogene Selbstwirksamkeitserwartung" - Fuchs & Schwarzer, 1994; "Weight Efficacy Life-Style Questionnaire (WEL)" - Clark et al., 1991; "SF 36 - Fragebogen zum Gesundheitszustand" - Bullinger und Kirchberger, 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Rader, Mag.a, Principal Investigator — FEM Süd
Locations (1):
- FEM Süd, Vienna, Austria

REFERENCES:
- See also: Homepage of the project (German) — http://www.rundum-gsund.at